CLINICAL TRIAL: NCT06956105
Title: A Randomized, Double-blind Sham-controlled Clinical Trial to Evaluate The Efficacy of Electrical Vestibular Stimulation (VeNS), Compared to a Sham Control For The Management Of Anxiety in Adolescents - The Modius Calm Adolescent Study
Brief Title: Electrical Vestibular Nerve Stimulation (VeNS) as a Treatment for Anxiety in Adolescents
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Neurovalens Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NV-MC-2025-001
Record Dates: First submitted 2025-04-23; First posted 2025-05-02 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: General Anxiety Disorder
MeSH Terms: conditions — Generalized Anxiety Disorder

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active VeNS device (Experimental): The active device utilizes a technology termed vestibular nerve stimulation (VeNS). The device will be placed on the head in a manner analogous to headphones and will deliver a small electrical current to the skin behind the ears, over the mastoid processes. Participants will be advised to use the device at home for 30 minutes per day.
  Interventions: Device: Modius Calm
- Sham device (Sham Comparator): The sham device looks identical to the active device. It will apply some stimulation to a user for a limited period of time (30 seconds), before tapering down to zero over a further 20 seconds, thus creating the impression of an active device. The device will be placed on the head in a manner analogous to headphones with hydrogel electrodes placed over the mastoid processes. Participants will be advised to use the device at home for 30 minutes per day.
  Interventions: Device: Sham device

INTERVENTIONS:
Device: Modius Calm — The Modius Calm device is a transdermal neurostimulation product. It consists of a battery-powered headset designed to deliver low-level energy in the form of a neurostimulation waveform that modulates the activity of the vestibular cranial nerve. The active Modius Calm device utilizes a technology called electrical vestibular nerve stimulation (VeNS). In the envisaged configuration the device will be placed on the head in a manner analogous to headphones and will deliver a small electrical current (a maximum of 1.5mA) to the skin behind the ears over the mastoid processes.
  Arms: Active VeNS device
Device: Sham device — The sham device is identical in appearance. The Modius Calm sham device follows this pattern by applying some stimulation to a user for a limited period of time (30 seconds), before tapering down to zero over a further 20 seconds, thus creating the impression of an active device.
  Arms: Sham device

SUMMARY:
Trial title: A Randomized, Double-blind Sham-controlled Clinical Trial to Evaluate The Efficacy of Electrical Vestibular Stimulation (VeNS), Compared to a Sham Control For The Management Of Anxiety in Adolescents - The Modius Calm Adolescent Study

The aim of this study: This investigation aims to evaluate the effects of VeNS for the treatment of Generalized Anxiety Disorder, to contribute to the field of knowledge about the neurological mechanisms to determine whether the relatively inexpensive, and non-invasive technique of VeNS can reduce the severity of GAD symptoms in adolescents.

Allocation: Randomized to either active device or control device usage.

Endpoint classification: Efficacy Study

Intervention Model: Parallel Assignment in 1:1 active to control allocation

Sample size: The aim is to recruit a total of up to 60 participants. The study will last 12 weeks in total for each subject.

DETAILED DESCRIPTION:
This double blind randomized controlled trial will enroll up to 60 subjects and will be conducted at the BGS MCH Hospital. The study will be randomized for a 8-week period with a 1:1 active to sham device allocation. Each participant will complete 5 stimulation sessions per week under the supervision of a researcher at the clinic. Each session will be 30 minutes on the day of usage. The scheduled study events are to be undertaken at the following timepoints:

* Baseline: Study Visit 1 (0-week timepoint for enrolment)
* Study Visit 2 (2-week timepoint)
* End of Study (4-week timepoint)
* Post-intervention follow-up at 2 weeks (6-week timepoint)
* Post-intervention follow-up at 6 weeks (10-week timepoint)
* Post-intervention follow-up at 8 weeks (12-week timepoint)

ELIGIBILITY:
Inclusion Criteria:

1. Signed Informed Consent
2. Signed Assent Form
3. Male or female, age ≥ 12 years and ≤ 17 years at the time of signing informed consent
4. GAD-7 score of >/=10 at screening
5. Can speak and read English
6. Ability and willingness to travel to the clinic to complete all study visits, stimulation sessions and procedures
7. Ability and willingness to adhere to 30 minutes usage of the device 5 days per week for the duration of the trial at clinic
8. Agree not to undergo any extreme lifestyle changes during the duration of the study that could impact anxiety e.g. dietary or exercise changes

Exclusion Criteria:

1. GAD-7 score of < 10 at screening
2. Medication for anxiety
3. Starting a new antidepressant during the study, or on an unstable dose of antidepressants within 3 months of starting study
4. Risk of persistent self-harm or suicide
5. Diagnosis or history of bipolar disorder
6. History of a current psychotic disorder such as schizophrenia or other non-mood disorder psychosis
7. Diagnosis of substance use disorder or dependence
8. Use of recreational drugs (e.g nalgesics, depressants, stimulants, and hallucinogens). Subject can enrol after a washout period of 30 days
9. History of diagnosed cognitive impairment / disorder such as delirium or dementia
10. Previous diagnosis of a chronic viral infection, for example hepatitis or HIV.
11. History of stroke or head injury requiring intensive care or neurosurgery
12. Presence of permanently implanted battery-powered medical device or stimulator (e.g., pacemaker, implanted defibrillator, deep brain stimulator, vagal nerve stimulator, etc.)
13. History of epilepsy
14. History of severe tinnitus or vertigo
15. History of skin breakdown, eczema or other dermatological condition (e.g. psoriasis) affecting the skin behind the ears.
16. History or presence of malignancy within the last year (except basal and squamous cell skin cancer and in-situ carcinomas)
17. History of vestibular dysfunction or another inner ear disease
18. Regular use (more than twice a month) of antihistamine medication within the last 6 months
19. Diagnosis of active migraines
20. Previous use of Modius device or any VeNS device
21. Participation in other clinical trials sponsored by Neurovalens
22. Any other medical condition, or medication use, that in the opinion of the PI is likely to make the subject refractory to VeNS.
23. Failure to use device daily during trial participation (no more than 7 consecutive days usage drop without reasonable explanation)

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2025-09-08 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
The change in GAD-7 score from baseline to 4 weeks | The GAD-7 shall be completed at baseline, 4 weeks (end of intervention) and 2 weeks, 6 weeks and 8 weeks post intervention .
  Generalized Anxiety Disorder 7 is a self-reported questionnaire for screening and severity measuring of generalized anxiety disorder. GAD-7 has seven items, which measure severity of various signs of GAD according to reported response categories with assigned points. The GAD-7 items include: 1) nervousness; 2) inability to stop worrying; 3) excessive worry; 4) restlessness; 5) difficulty in relaxing; 6) easy irritation; and 7 fear of something awful happening. Scores of 5, 10, and 15 are taken as the cut-off points for mild, moderate and severe anxiety, respectively. The GAD-7 was originally validated in a primary care sample and a cut-off score of 10 had a sensitivity value of 0.89 and a specificity value of 0.82 for identifying GAD.

SECONDARY OUTCOMES:
Change in the Insomnia Severity Index (ISI) score from baseline to 4 weeks | The ISI shall be completed at baseline and repeated at both 2 (mid-point) and 4 weeks (end of study).
  The Insomnia Severity Index (ISI) is a validated short, self-report screening assessment tool designed to evaluate insomnia by measuring an individual's perception of both day and night symptoms of insomnia. The Index consists of seven items which are each assessed in terms of perceived difficulty: falling sleep, staying asleep, and time of awakening, satisfaction with current sleep pattern, interference with daily functioning, noticeability by others of impact of lack of sleep, and degree of perceived distress or concern caused by the sleep problem.
Change in the Mental Health-related Quality of Life (SF-36) mental component (MC) score from baseline to 4 weeks | The SF-36 will be administered at baseline, mid-point (2 weeks), and end of study (4 weeks).
  The SF-36 is a widely used, self-reported health-related quality of life (HRQoL) questionnaire designed to measure functional health and well-being from the patient's perspective. It assesses eight key domains: physical functioning, role limitations due to physical health, bodily pain, general health perceptions, vitality (energy/fatigue), social functioning, role limitations due to emotional problems, and mental health. Each domain is scored individually and can be combined into two overall summary scores: the Physical Component Summary (PCS) and the Mental Component Summary (MCS). In this study, the PCS and MCS scores will be the primary focus, allowing to evaluate changes in both physical and mental aspects of health over time. The questionnaire has been validated in diverse populations, including adolescents, and is commonly used in clinical trials and health outcome research.
Change in the Physical Health-related Quality of Life (SF-36) physical component (MC) score from baseline to 4 weeks. | The SF-36 will be administered at baseline, mid-point (2 weeks), and end of study (4 weeks).
  The SF-36 is a widely used, self-reported health-related quality of life (HRQoL) questionnaire designed to measure functional health and well-being from the patient's perspective. It assesses eight key domains: physical functioning, role limitations due to physical health, bodily pain, general health perceptions, vitality (energy/fatigue), social functioning, role limitations due to emotional problems, and mental health. Each domain is scored individually and can be combined into two overall summary scores: the Physical Component Summary (PCS) and the Mental Component Summary (MCS). In this study, the PCS and MCS scores will be the primary focus, allowing to evaluate changes in both physical and mental aspects of health over time. The questionnaire has been validated in diverse populations, including adolescents, and is commonly used in clinical trials and health outcome research.

CONTACTS AND LOCATIONS:
Overall Officials: Sai Sailesh Kumar Goothy, Principal Investigator — BGS MCH Hospital
Locations (1):
- BGS MCH Hospital, Bangalore, India

IPD SHARING:
Plan to Share IPD: No